CLINICAL TRIAL: NCT06310642
Title: A Prospective Single-Blinded Randomized Field-Based Trial to Evaluate the Prophylactic Treatment of Oral Prochlorperazine for Acute Mountain Sickness
Brief Title: Efficacy of Prophylactic Treatment of Oral Prochlorperazine for Acute Mountain Sickness
Acronym: PAMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Peter Richman, MD, Professor and Research Director, Department of Emergency Medicine, CHRISTUS Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-217
Record Dates: First submitted 2024-01-08; First posted 2024-03-15 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: AMS; Acute Mountain Sickness
Keywords: Prochlorperazine; AMS; LLAMS Score; Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Diphenhydramine; Prochlorperazine

STUDY DESIGN:
Intervention Model Description: Enrolled a cohort of consenting, healthy subjects aged >17 years. Thirty subjects enrolled in the study. 15 subjects received prochlorperazine. 15 subjects received placebo.
Who Masked: Participant
Masking Description: Patients were blinded in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prochlorperazine 10 mg (Experimental): Subjects received 10 mg Prochlorperazine one time.
  Interventions: Other: Immediate descent from altitude.; Drug: Diphenhydramine; Drug: Prochlorperazine 10 mg
- Placebo (Placebo Comparator): Subjects received Placebo one time.
  Interventions: Other: Immediate descent from altitude.; Drug: Diphenhydramine

INTERVENTIONS:
Other: Immediate descent from altitude. — Immediate descent from altitude for severe symptoms or anyone who wished to discontinue their participation in the study.
Drug: Diphenhydramine — Diphenhydramine was available to counteract any potential extrapyramidal side effects of the study drug. The use of Diphenhydramine for this purpose is well established.
  Other Names: Benadryl
Drug: Prochlorperazine 10 mg — Subjects in the Prochlorperazine arm were administered 10mg PO Prochlorperazine immediately prior to ascent
  Arms: Prochlorperazine 10 mg

SUMMARY:
A field-based trial was conducted to determine if oral prochlorperazine demonstrates efficacy in the prophylactic treatment of AMS, and/or decreases the incidence of the symptoms of acute mountain sickness including headache, GI symptoms, fatigue and dizziness based on data collected in the Lake Louise AMS score.

DETAILED DESCRIPTION:
This was a prospective, single-blinded, field-based interventional trial involving consenting, healthy subjects aged >17 years. The study was conducted on the big Island of Hawaii, at sea level and at the summit of Mauna Kea volcano. Following randomization, subjects received either placebo or 10mg prochlorperazine, then immediately drove for 2 hours from sea level to the volcano summit (4205m). Participants spent 240 min at the summit, and they recorded their symptoms. AMS was defined by the previously validated Lake Louise Acute Mountain Sickness Score (LLAMS). Categorical variables were analyzed by chi-square; continuous variables analyzed by t-tests.

ELIGIBILITY:
Inclusion Criteria - Healthy subjects aged >17 years

Exclusion criteria-subject meets any of the following:

* Known allergy or contraindication to the study drug.
* Known or suspected pregnancy.
* Use of another analgesic or antiemetic within 8 hours of enrollment.
* History of chronic headaches.
* Inability to provide informed consent.
* Use of central nervous system depressants, including alcohol, opiates, and/or barbiturates, within 24 hours of the study start time.
* History of severe depression.
* History of dementia.
* Prior ascent and stay at 2500m for duration over 6 weeks within 30 days prior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Mean Lake Louise Acute Mountain Sickness Score (LLAMS) was utilized to compare symptoms of acute mountain sickness between the prochlorperazine and placebo groups | LLAMS Scores were recorded 360 minutes post study drug administration (which equals 120 minutes of driving time to the summit and an additional 240 minutes spent at the summit)
  The study drug was administered at sea level (time 0). Immediately thereafter, participants drove 120 minutes to the summit. They spent an additional 240 minutes at the summit. Symptoms were recorded 360 minutes after drug administration while still at the summit. The primary outcome was the difference in mean LLAMS scores between the prochlorperazine and placebo groups (t-tests).
  Previously validated Lake Louise Acute Mountain Sickness Score (LLAMS) were utilized. Categorical variables were analyzed by chi-square; continuous variables analyzed by t-tests.

SECONDARY OUTCOMES:
Subjects meeting Lake Louise Acute Mountain Sickness Score (LLAMS) criteria for acute mountain sickness between the prochlorperazine and placebo groups | LLAMS Scores were recorded 360 minutes post study drug administration (which equals 120 minutes of driving time to the summit and an additional 240 minutes spent at the summit)
  The study drug was administered at sea level (time 0). Immediately thereafter, participants drove 120 minutes to the summit. They spent an additional 240 minutes at the summit. Symptoms were recorded 360 minutes after drug administration while still at the summit. Acute mountain sickness defined as having a headache score of at least one point, and a total score of at least three points. The prochlorperazine and placebo groups were compared for incidence of acute mountain sickness (chi-square)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Richman, MD, Principal Investigator — CHRISTUS Health
Locations (1):
- CHRISTUS Health-Texas A&M Spohn Emergency Medicine Residency, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan.

REFERENCES:
- [Background] Smedley T, Grocott MP. Acute high-altitude illness: a clinically orientated review. Br J Pain. 2013 May;7(2):85-94. doi: 10.1177/2049463713489539. PMID 26516505
- [Background] Klocke DL, Decker WW, Stepanek J. Altitude-related illnesses. Mayo Clin Proc. 1998 Oct;73(10):988-92; quiz 992-3. doi: 10.4065/73.10.988. PMID 9787751
- [Background] Irons HR, Salas RN, Bhai SF, Gregorie WD, Harris NS. Prospective Double-Blinded Randomized Field-Based Clinical Trial of Metoclopramide and Ibuprofen for the Treatment of High Altitude Headache and Acute Mountain Sickness. Wilderness Environ Med. 2020 Mar;31(1):38-43. doi: 10.1016/j.wem.2019.11.005. Epub 2020 Feb 11. PMID 32057631
- [Background] Luks AM, Auerbach PS, Freer L, Grissom CK, Keyes LE, McIntosh SE, Rodway GW, Schoene RB, Zafren K, Hackett PH. Wilderness Medical Society Clinical Practice Guidelines for the Prevention and Treatment of Acute Altitude Illness: 2019 Update. Wilderness Environ Med. 2019 Dec;30(4S):S3-S18. doi: 10.1016/j.wem.2019.04.006. Epub 2019 Jun 24. PMID 31248818
- [Background] Netzer N, Strohl K, Faulhaber M, Gatterer H, Burtscher M. Hypoxia-related altitude illnesses. J Travel Med. 2013 Jul-Aug;20(4):247-55. doi: 10.1111/jtm.12017. Epub 2013 Mar 11. PMID 23809076
- [Background] Lu H, Wang R, Xiong J, Xie H, Kayser B, Jia ZP. In search for better pharmacological prophylaxis for acute mountain sickness: looking in other directions. Acta Physiol (Oxf). 2015 May;214(1):51-62. doi: 10.1111/apha.12490. Epub 2015 Mar 28. PMID 25778288
- [Background] Kanaan NC, Peterson AL, Pun M, Holck PS, Starling J, Basyal B, Freeman TF, Gehner JR, Keyes L, Levin DR, O'Leary CJ, Stuart KE, Thapa GB, Tiwari A, Velgersdyk JL, Zafren K, Basnyat B. Prophylactic Acetaminophen or Ibuprofen Results in Equivalent Acute Mountain Sickness Incidence at High Altitude: A Prospective Randomized Trial. Wilderness Environ Med. 2017 Jun;28(2):72-78. doi: 10.1016/j.wem.2016.12.011. Epub 2017 May 4. PMID 28479001
- [Background] Olson LG, Hensley MJ, Saunders NA. The effects of combined morphine and prochlorperazine on ventilatory control in humans. Am Rev Respir Dis. 1986 Apr;133(4):558-61. doi: 10.1164/arrd.1986.133.4.558. PMID 3963624